CLINICAL TRIAL: NCT01731743
Title: Evaluation of Visual Acuity and Patient Satisfaction With AT LISA TRI 839MP Intraocular Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carl Zeiss Meditec AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 839 MP HEN 402-11
Record Dates: First submitted 2012-11-19; First posted 2012-11-22 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- implantation of a trifocal IOL (AT LISA tri 839MP) (Other)
  Interventions: Device: AT LISA tri 839MP

INTERVENTIONS:
Device: AT LISA tri 839MP

SUMMARY:
The purpose of the study is to evaluate the far, intermediate and near visual acuities with a trifocal IOL.

DETAILED DESCRIPTION:
After bilateral cataract surgery, monocular and binocular uncorrected (UCVA) and best distance corrected visual acuity (BCVA) will be measured at far (4m), intermediate (80 cm) and near (40 cm) distance as well as the subjective refraction.

A patient questionnaire will be used to assess the patient satisfaction and spectacle independence.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman, over 50 years of age
* Bilateral implantation of a trifocal intraocular lens
* Capsular bag implantation

Exclusion Criteria:

* Existing ocular pathology
* Surgical complications
* Corneal astigmatism ≥ 1.0D

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2012-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Intermediate visual acuity | up to 3 months postoperatively
  Monocular and binocular uncorrected and best distance corrected

SECONDARY OUTCOMES:
near and far visual acuity | 1 and 3 month postoperatively
  Monocular and binocular uncorrected and best distance corrected

OTHER OUTCOMES:
Patient satisfaction and spectacle independence | 1 and 3 month postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Carl Zeiss Meditec AG, Berlin, Germany